CLINICAL TRIAL: NCT01649024
Title: A Second-line, Single Arm, Phase II Clinical Study With Tremelimumab, a Fully Human Anti-CTLA-4 Monoclonal Antibody as Monotherapy in Patients With Unresectable Malignant Mesothelioma
Brief Title: A Clinical Study With Tremelimumab as Monotherapy in Malignant Mesothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Responsible Party: Principal Investigator, Michele Maio, Head of Medical Oncology and Immunotherapy, University Hospital of Siena, Azienda Ospedaliera Universitaria Senese
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MESOT-TREM-2008; 2008-005171-95 (EudraCT Number)
Record Dates: First submitted 2012-07-18; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Malignant Mesothelioma
Keywords: Tremelimumab; Malignant Mesothelioma; anti-CTLA-4 mAb
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm of Tremelimumab (Experimental): Tremelimumab is administered at 15 mg/kg on day 1 every 12 weeks for 4 doses
  Interventions: Drug: Tremelimumab

INTERVENTIONS:
Drug: Tremelimumab — Given IV
  Other Names: CP-675,206

SUMMARY:
The study is designed to define the immunologic and clinical activity of Tremelimumab in patients with advanced mesothelioma.

DETAILED DESCRIPTION:
No effective standard treatment can improve significantly the prognosis of malignant mesothelioma (MM) patients. However, there is evidence that MM patients may benefit from immunotherapeutic agents.

Clinical studies examining CTLA-4 blockade are providing convincing evidences on the immunobiological effects and on the clinical activity of this new class of immunomodulating therapeutic agents, likely due to their ability to stimulate patients'immune system to more effectively attack tumor cells by blocking a negative regulatory signal.

Tremelimumab is a fully human anti-CTLA-4 monoclonal antibody (mAb), developed as an IgG2 isotype to minimize complement activation and reduce the risk of cytokine storm. As a single agent, Tremelimumab can induce durable tumor regression in 7-10% of patients with advanced melanoma. Tremelimumab has been tested in several clinical trials as single-agent or in combination with other agents in different solid tumors.

The evidences above unveil a strong immunologic potential of treatment with Tremelimumab also in MM patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant mesothelioma (MM)
* Have received only one prior systemic chemotherapy platinum-based regimen for advanced MM
* Disease not amenable to curative surgery
* No known brain metastasis
* Age 18 and over
* Performance status 0-2
* Life expectancy > 12 weeks
* Adequate hematologic, hepatic and renal function
* Not pregnant or nursing
* Patient must be willing and able to provide written informed consent, and the trial have to be approved by the institutional review board at each institution

Exclusion Criteria:

* Symptomatic chronic inflammatory or autoimmune disease
* Active hepatitis B or C
* Clinically relevant cardiovascular disease, i.e., myocardial infarction or other severe coronary artery diseases within the prior 6 months, cardiac arrythmia requiring medication, uncontrolled hypertension, overt cardiac failure or not compensated chronic heart disease in NYHA class II or more
* History of psychiatric disabilities, potentially interfering with the capability of giving adequate informed consent
* Uncontrolled active infections
* Other concurrent chemotherapy, immunotherapy, radiotherapy or investigational agents
* History of other malignancies except for adequately treated basal cell carcinoma or squamous cell skin cancer or carcinoma of cervix, unless the patient has been disease-free for at least 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response by modified Response Evaluation Criteria in Solid Tumor (RECIST) | Weeks 24
  The objective tumor response is defined as a confirmed complete response (CR) or partial response (PR) according to the modified RECIST criteria for pleural mesothelioma

SECONDARY OUTCOMES:
Disease control rate | 1 year
  Disease control rate (DCR) is the proportion of treated subjects that achieved confirmed complete response, or partial response, or stable disease.
  The DCR is assessed using the modified RECIST criteria for pleural mesothelioma
Progression free survival | 1 year
  Progression free survival is computed from the first day of study treatment to the day of documented progression according to the modified RECIST criteria for pleural mesothelioma or death, whichever occurs first
Safety | 2 years
  The assessment of safety includes serious and non-serious adverse events according to NCI-CTC criteria version 3.0. In addition, laboratory evaluation, abnormal vital signs and physical examination findings are also included.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Maio, MD, Principal Investigator — Medical Oncology and Immunotherapy Unit, University Hospital of Siena
Locations (1):
- Medical Oncology and Immunotherapy Unit, University Hospital of Siena, Siena, Italy

REFERENCES:
- [Derived] Calabro L, Morra A, Fonsatti E, Cutaia O, Amato G, Giannarelli D, Di Giacomo AM, Danielli R, Altomonte M, Mutti L, Maio M. Tremelimumab for patients with chemotherapy-resistant advanced malignant mesothelioma: an open-label, single-arm, phase 2 trial. Lancet Oncol. 2013 Oct;14(11):1104-1111. doi: 10.1016/S1470-2045(13)70381-4. Epub 2013 Sep 11. PMID 24035405